CLINICAL TRIAL: NCT01112696
Title: An Inpatient Performance Evaluation of a New Subcutaneous Glucose Sensor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CEP 221
Record Dates: First submitted 2010-04-27; First posted 2010-04-28 (Estimated); Results first posted 2012-08-27 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2017-12

CONDITIONS: Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus
Keywords: diabetes; glucose sensor; CGM
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sensor (Other): All subjects that wear sensors (all subjects)
  Interventions: Device: Sensor wear

INTERVENTIONS:
Device: Sensor wear — All subjects to wear sensors
  Other Names: Enlite Sensor

SUMMARY:
The purpose of the study is to assess the performance of a new subcutaneous glucose sensor over a seven-day sensor life when used with currently marketed Medtronic Diabetes devices. In addition performance will be calculated for use of the new sensor with proposed new devices using new calibration algorithms.

DETAILED DESCRIPTION:
The first generation Medtronic MiniMed Subcutaneous Glucose Sensor (Sof-Sensor) was originally approved by the FDA for commercialization as part of the Continuous Glucose Monitoring System (CGMS) on June 15, 1999 (PMA 980022). The Sensor is composed of a microelectrode with a thin coating of glucose oxidase beneath several layers of biocompatible membrane. This same sensor was used as part of subsequent continuous glucose monitoring (CGM) systems, such as the Guardian REAL-Time and Paradigm REAL-Time sensor augmented insulin pump. The current configuration of sensor has undergone in vitro and in vivo testing. A new second-generation glucose sensor (herein referred to as the Comfort Sensor) has been developed. The first-generation glucose sensor was approved with reported sensor accuracy (MAD) of 18%; it was labeled for a maximum use duration of 72 hours, using only the abdomen as an insertion site. The new sensor is shorter and has a smaller diameter, with a smaller gauge introducer needle. The new sensor inserter is designed to be used with the new sensor. The objectives of this study are to 1) Assess performance of the Comfort Sensor when used over a period of seven days with currently available devices, and 2) Assess performance of the Comfort Sensor when used over a period of seven days using new calibration algorithms (post-processed with algorithm for future devices). Accuracy data will be calculated based on comparing calibrated glucose sensor values to a "gold standard" (YSI plasma glucose values) in adult subjects during in-clinic testing, and on comparing calibrated glucose sensor values to glucose meter values during in-home testing. The devices that will be used for gathering sensor data during this study will be: 1) the Comfort Sensor, 2) the MiniLink (Transmitter), 3) the Guardian REAL-Time Display Device and 4) the CGMS iPro.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18 through 75 inclusive
2. Diagnosed with Type 1 or type 2 Diabetes Mellitus, using insulin to treat their diabetes (Each site's and overall study enrollment of subjects with Type 2 diabetes will target 20% of the total number)
3. Willingness to perform required study and data collection procedures and to adhere to operating requirements of the Guardian REAL-TIME and CGMS iPro Systems
4. Willingness to perform at least 4 capillary blood glucose tests per day while wearing the Guardian REAL-TIME and CGMS iPro Systems
5. Willingness to participate in a 10 hour frequent blood sampling session during the study
6. Subject agrees to comply with the study protocol requirements
7. Informed Consent, HIPAA Authorization, and California Experimental Subject Bill of Rights (if applicable) signed by the subject
8. The Subject is willing to wear both the Guardian REAL-Time and CGMS iPro Systems for 14 days (~340 hours)

Exclusion Criteria:

1. The Subject has a history of tape allergies that have not been resolved
2. The Subject has any skin abnormality (e.g. psoriasis, rash, staphylococcus infection) that has not been resolved and would inhibit them from wearing the sensors
3. Any additional condition(s) that in the Investigator's opinion would warrant exclusion from the study or prevent the Subject from completing the study
4. Subject is currently participating in an investigational study (drug or device)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-04; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Lee, MD, Study Director — Medtronic Diabetes
Locations (3):
- United States (3):
  - AMCR Institute, Inc., Escondido, California
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - Rainier Clinical Research Center, Inc., Renton, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Sensor Users (All Subjects)
Period: Overall Study
Arm/Group | Group 1
Started | 100
Completed | 98
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Group 1
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 92
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 69
Region of Enrollment [Number; unit: participants]
  United States | 100

OUTCOME MEASURES:

1. Primary Outcome: Glucose Sensor Accuracy When Compared to Laboratory Standard (YSI): Proportion of Glucose Sensor Readings That Met Accuracy Criteria
Description: The primary accuracy parameter (primary effectiveness endpoint) was the comparative readings of paired sensor and YSI glucose readings, measured on days 1 through 6. Accuracy is defined as within 20% agreement between YSI and paired sensor (within 20 mg/dL if YSI <80 mg/dL). Accuracy ranges from 0 - 100, with higher number suggests better accuracy.
Time Frame: Days one through six of sensor use
Population: 98 subjects of 100 enrolled subjects (a total of 5857 paired sensor and YSI readings) completed participation in the inpatient frequent blood sampling procedure.
Measure: Number (95% Confidence Interval); unit: paired sensor and YSI glucose readings
Units Other Than Participants: paired YSI/sensor glucose values
Groups:
- All Completed Subjects: All subjects that completed the frequent blood sampling procedure
Arm/Group | All Completed Subjects
Number analyzed (Participants) | 98
Number analyzed (paired YSI/sensor glucose values) | 5857
paired sensor and YSI glucose readings | 79.45 [75.93 to 82.96]

2. Secondary Outcome: Device Related Moderate or Device Related Severe Adverse Events
Description: Device related moderate adverse event: low level of inconvenience or concern to the subject and may interfere with daily activities but is usually improved by simple therapeutic remedy.
  Device related severe adverse event: interrupts a subject's daily activity and typically requires intervening treatment.
  Note: device related determination is made by the site that there is a reasonable possibility that the adverse event may have been caused by the device.
Time Frame: days one through six of sensor wear
Measure: Count of Participants; unit: Participants
Arm/Group | Sensor
Number analyzed (Participants) | 100
Participants | 0

ADVERSE EVENTS:
Arm/Group | Group 1
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less